CLINICAL TRIAL: NCT06931691
Title: A Multi-center, Ambispective Cohort Study to Evaluate the Impact of Iptacopan on Disease Management, Treatment-Related Outcomes and Healthcare Resource Utilization for Adult Patients With Paroxysmal Nocturnal Hemoglobinuria in China
Brief Title: A Multi-center, Ambispective Cohort Study to Evaluate the Impact of Iptacopan for Adult Patients With PNH in China
Acronym: PNH-NIS
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023C1CN01
Record Dates: First submitted 2025-03-14; First posted 2025-04-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Phase IV; Adult Patients; Paroxysmal Nocturnal Hemoglobinuria; LNP023
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort1: PNH patients with a confirmed diagnosis of PNH in the medical record and who had never received complement inhibitor therapy (complement inhibitor naive patients)
  Interventions: Drug: LNP023
- Cohort 2: PNH patients with a confirmed diagnosis of PNH in the medical record who had been treated with a stable dose of a C5 complement inhibitor (e.g., eculizumab) for at least 3 months (C5i-treated patients; this cohort will be only start enrollment after the indication for iptacopan is to be approved in China).
  Interventions: Drug: LNP023

INTERVENTIONS:
Drug: LNP023 — Capsules for oral administration
  Other Names: Iptacopan Hydrochloride

SUMMARY:
The implementation of new standards for the management of PNH and the use of iptacopan in patients with PNH are expected to change the treatment landscape and improve the overall prognosis of patients.

Based on these backgrounds, we plan to conduct a real-world study of iptacopan to further evaluate its impact on treatment-related outcomes, disease management, and healthcare resource utilization in Chinese patients with PNH.

ELIGIBILITY:
Inclusion criteria For Cohort 1,

Patient who meets all the following criteria can be included in this study:

1. Age ≥ 18 years at the time of signing the ICF;
2. Patient with a documented diagnosis of PNH;
3. Patient who has never received complement inhibitor therapy;
4. Patient who is initiating iptacopan therapy; Patient who is initiating iptacopan therapy must start the first dose within 60 days of signing the ICF;
5. Documented vaccination against Neisseria meningitidis and Streptococcus pneumoniae and the date of vaccination must be at least 2 weeks prior to the date of iptacopan initiation; If an urgent prescription for Iptacopan is needed, it is recommended that the antibiotic be used continuously according to the drug label until 14 days after the vaccination is completed, and that the vaccination be completed as soon as possible.
6. Patient who has signed the ICF.

For Cohort 2,

Patient who meets all the following criteria can be included in this study:

1. Age ≥ 18 years at the time of signing the ICF;
2. Patient with a documented diagnosis of PNH; Patients who have been receiving stable treatment with C5 complement inhibitors for at least three months prior to enrollment;
3. Patient who is initiating iptacopan therapy; Patient who is initiating iptacopan therapy must start the first dose within 60 days of signing the ICF;
4. Documented vaccination against Neisseria meningitidis and Streptococcus pneumoniae and the date of vaccination must be at least 2 weeks prior to the date of iptacopan initiation;
5. If an urgent prescription for Iptacopan is needed, it is recommended that the antibiotic be used continuously according to the drug label until 14 days after the vaccination is completed, and that the vaccination be completed as soon as possible.
6. Patient who has signed the ICF. Exclusion criteria

For Cohort 1 and Cohort 2, patients who meet any of the following criteria will meet the exclusion criteria for this study:

1. Participating in an interventional PNH clinical study;
2. Have an active systemic bacterial, viral (incl. COVID-19) or fungal infection within 14 days prior to first dose;
3. Documented with a history of recurrent invasive infections, e.g. active systemic bacterial, viral or fungal infection within 14 days prior to first dose;
4. Documented with a history of HIV infection;
5. Women who are pregnant or breastfeeding or intending to conceive during the study period;
6. Existence of bone marrow failure (reticulocytes < 100 × 109/L, platelets < 30 × 109/L, and neutrophils < 0.5 × 109/L) determined by the investigator;
7. Other conditions that are not suitable for participating in the study, in the judgment of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult PNH patients receiving iptacopan for the first time, including those who are complement inhibitor naive and treated
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-04-20 (Estimated); Study Completion 2027-04-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin (Hb) levels at designated time points | Baseline, 12 months
  Assessment of the Hematological Response to iptacopan.

SECONDARY OUTCOMES:
Number of participants having Hb normalization (Hb level ≥ 12 g/dL) after iptacopan initiation. | 12 months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Duration of Hb level ≥ 12 g/dL within a 12-month | 12 months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Change from baseline in LDH Levels after iptacopan initiation | Baseline, 12 Months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Number of participants with LDH levels ≤ 1.5 x ULN before vs. after iptacopan initiation | 12 months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Number of participants having LDH normalization before and after iptacopan initiation | 12 monhts
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Duration of LDH level ≤ 1.5 x ULN within 12 months | 12 months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Change from baseline in ARC Levels after iptacopan initiation | Baseline, 12 monhts
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Number of participants having ARC normalization before and after iptacopan initiation | Baseline, 12 months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Change from baseline in bilirubin after iptacopan initiation | Baseline, 12 months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Number of participants with hepatosplenomegaly before and after iptacopan initiation | Baseline, 12 months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Number of participants with a positive coomb's test after iptacopan initiation | 12 months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Number of participants with PNH related signs or symptoms before and after iptacopan treatment | Baseline, 12 months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Change from baseline in PNH clone value | Baseline, 12 months
  Change from baseline in flow cytometry results to assess the impact of iptacopan on Treatment-Related Outcomes.
Rate, reasons (complement activation conditions (CAC), missed doses, etc.), duration, and interventions for breakthrough hemolysis (BTH) | 12 months
  Assessing the Impact of iptacopan on Treatment-Related Outcomes
Change from baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale after iptacopan initiation | Baseline, 12 months
  FACIT is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function to assess the Impact of iptacopan on Treatment-Related Outcomes. The minimum value is 0 and maximum value is 52, and higher scores mean a worse outcome.
Work Productivity and Activity Impairment Questionnaire-Specific Health Problems (WPAI-SHP) at each visit, change from baseline in WPAI-SHP after iptacopan initiation | Baseline, 12 months
  WPAI-SHP is a tool used to measure the impact of health problems on work productivity and regular activities. The scale includes several components.
  Absenteeism: This measures the percentage of work time missed due to a specific health problem.
  Presenteeism: This measures the percentage of impairment while working due to the health problem.
  Work productivity loss: This combines absenteeism and presenteeism to measure overall work impairment.
  Activity impairment: This measures the percentage of impairment in regular activities due to the health problem.
  The scores are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, which means worse outcomes.
Adverse events (AEs) and Serious adverse events (SAEs) occurring during treatment with iptacopan | 12 monhts
  Assessing the safety of iptacopan
Treatment regimen for PNH 12 months before iptacopan treatment; reasons of discontinuation of previous complement inhibitor; | Baseline
  Assessing the impact of iptacopan on disease management
Use of concomitant medications (e.g., corticosteroids, androgen, immunosuppressants, anti-coagulants, etc.) for PNH and PNH-related complications (e.g. thrombosis, renal failure, etc.) before and after iptacopan treatment; | Baseline, 12 months
  Assessing the impact of iptacopan on disease management
Duration of iptacopan treatment, reasons for discontinuation, switching to other treatments, proportion of patients who switch from iptacopan to other treatments; | 12 monhts
  Assessing the impact of iptacopan on disease management
Number of participants with blood transfusion before and after iptacopan treatment, duration and number of units of blood transfusion due to BTH | Baseline, 12 months
  Assessing the impact of iptacopan on disease management
Number of participants hospitalized, outpatient, emergency room and intensive care unit (ICU) visits related to PNH | 12 monhts
  Assessing the impact of iptacopan on healthcare resource utilization
Length of inpatient stay related to PNH | 12 months
  Assessing the impact of iptacopan on healthcare resource utilization

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Wuhan

IPD SHARING:
Plan to Share IPD: No